CLINICAL TRIAL: NCT04693611
Title: Prefrontal Cortex Dynamics of the Elderly During a Cognitive Stimulation Programme: A Randomized and Controlled Trial in Old Adults With Normal Cognition and Mild Cognitive Impairment
Brief Title: Prefrontal Cortex Dynamics of the Elderly During a Cognitive Stimulation Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEDIARA - Assoc. Solidariedade Social de Ribeira de Fráguas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16122020
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-02

CONDITIONS: Dementia; Neurocognitive Disorders; Cognitive Impairment; Cognitive Dysfunction; Cognitive Decline; Cognition Disorders in Old Age
Keywords: brain activity; mood; functional near-infrared spectroscopy; prefrontal cortex; older adults; cognitive stimulation
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who meet the inclusion criteria will be randomised to the CS intervention group or to the control group that will maintain their usual treatment.
  Participants in the intervention group will participate in two CS sessions per 12 weeks besides their treatment as usual.
  Interventions: Behavioral: Individual cognitive stimulation therapy (iCST); Procedure: Functional near-infrared spectroscopy (fNIRS)
- Control Group (No Intervention): Participants in the control group will maintain their usual treatment: social interaction activities, stimulation of personal skills, and any prescribed dementia-specific medication.

INTERVENTIONS:
Behavioral: Individual cognitive stimulation therapy (iCST) — The intervention group will receive 24 individual CS sessions per participant. Each session will last approximately 45 minutes and will have the following structure: session introduction (5 minutes); reality orientation (10 minutes); stimulation of cognitive domain (25 minutes); session closure (5 minutes). The sessions will be led by a previously trained therapist. The intervention program will include several activities based on the principles of CS and adjusted for participants without any neurocognitive disorder.
  Arms: Intervention Group
Procedure: Functional near-infrared spectroscopy (fNIRS) — The acquisition by fNIRS will be performed in each CS session in four regions of interest (ROIs) in the prefrontal cortex: left dorsolateral prefrontal cortex (LDLPFC); left medial prefrontal cortex (LMPFC); right medial prefrontal cortex (RMPFC); right dorsolateral prefrontal cortex (RDLPFC).
  Arms: Intervention Group

SUMMARY:
This research aims to evaluate the effect of cognitive stimulation (CS) on the functioning of the prefrontal cortex (PFC), seeking an analysis of both cerebral hemodynamics in neuroplasticity and aspects related to the initiation of neurodegenerative processes. The intervention presents an individual format and the participants are elderly without or with neurocognitive disorders (NCD). Concretely, to assess the effects of individual CS on global cognition, and mood, as well as to analyze neuronal activity with oxygenation, volume and blood flow in the brain, evaluating the impact of cognitive stimulation on brain hemodynamics. Participants in the intervention group receive two 45 min-session of CS per week for 12 weeks in addition to their treatment as usual. Participants in the control group will maintain their treatment as usual.

DETAILED DESCRIPTION:
Faced with an unprecedented global ageing population and the current COVID-19 pandemic, the risk of social vulnerability increases in the elderly population, promoting the development and aggravation of neurodegenerative diseases, in particular NCD. The diagnostic criteria for this pathology emphasizes cognitive changes, and as such is based clinically on cognitive decline.

The PFC is considered the centre of cognitive function, where it encompasses attention, memory and executive functions.

Attention is the cognitive function that allows us to orient to the relevant stimuli and process them to respond accordingly. Given its functionality, it is distinguished into three types of attention: selective, divided and sustained. Attentional dysfunction can be present in several conditions where cognitive deficit is the main symptom, such as Alzheimer's disease.

With regard to memory, it is subdivided according to time storage, i.e. short or long term. Short-term memory is capable of operating with certain perceived information for a limited space of time and can later be forgotten or transferred to long-term memory. Two other complementary components are distinguished in this type of memory: immediate memory and recent memory. Long-term memory is a latent memory with unlimited capacity that can remain outside the conscious circuit until circumstances require another mode of response. It involves separate, interdependent and dynamic processes of storage, consolidation and evocation. It is made up of two major subsystems: implicit or non-declarative memory, and explicit or declarative memory.

Regarding executive functions, they designate the cognitive processes of control and integration aimed at the execution of behaviour directed at complex objectives, requiring sub-components such as attention, programming, time sequencing, inhibition of competing processes and information, monitoring and selection of strategies. Executive functions include various processes such as working memory, planning, response to reactions and error corrections, cognitive flexibility, inhibition, decision making.

There is evidence that in the early stages of NCD, people are able to learn and improve their cognitive function through interventions such as CS. CS is recommended by the National Institute for Health and Clinical Excellence as a non-pharmacological therapy for people with mild to moderate NCD and is an intervention where the cognitive domains are not used in isolation but integrated. An individual format is associated with better results. In a systematic review on CS, studies have shown strong evidence that CS has a positive impact on cognitive function, depression, daily life activities and behaviour for people with NCD.

However, no studies are known that have analyzed prefrontal cortex activity in the elderly population associated with a functional method of infrared spectroscopy (fNIRS). This method provides information on hemodynamic changes associated with cortical activation by measuring in a non-invasive way changes in the relative ratios of deoxygenated hemoglobin (HHb) and oxygenated hemoglobin (HbO2).

Monitoring and recording the dynamics in the PFC of the elderly during a cognitive stimulation programme with the fNIRS method may contribute to expanding knowledge about aspects related to neurodegenerative processes and cognitive function in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older.
* Being able to communicate and understand.
* Being a native Portuguese speaker.
* Educational level equal to or higher than 4 years old.
* Have given informed consent for the project, duly completed and signed, after prior information.
* Have a score of 22 or more points in the MMSE.

Exclusion Criteria:

* Suffering from an acute or severe illness that prevent participation in the intervention sessions.
* Severe sensory and physical limitations that prevent participation.
* Low level of consciousness and minimal attention span.
* Presence of severe neuropsychiatric symptoms (such as agitation, psychosis, severe depressive and anxiety symptoms, apathy), or presence of uncontrolled delirium that would prevent participation in the sessions.
* History of seizures or cerebrovascular disease.
* Movement disorders diagnosis.
* Psychoactive substances consumption.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Mini-Mental State Examination (MMSE) | baseline
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. MMSE is a brief cognitive screening test. Scores range between 0-30 points. Higher scores indicate better cognitive function.
Change in cognitive functioning evaluated through MMSE | 12 weeks after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. MMSE is a brief cognitive screening test. Scores range between 0-30 points. Higher scores indicate better cognitive function.
Executive functions evaluated through Frontal Assessment Battery (FAB) | baseline
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points. Higher scores indicate better cognitive function.
Change in executive functions evaluated through FAB | 12 weeks after the beginning of the intervention
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and postintervention assessment. FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points. Higher scores indicate better cognitive function.
Prefrontal cortex activation pattern through a fNIRS | baseline
  Analysis of Oxyhemoglobin (HbO2) and Deoxyhemoglobin (HHb) variation in four regions of interest (ROIs) in the PFC: left prefrontal dorsolateral cortex (LDLPFC); left medial prefrontal cortex (LMPFC); right medial prefrontal cortex (RMPFC); right dorsolateral prefrontal cortex (RDLPFC). An increase in brain activity is generally assumed to reflect an increase in HbO2 and decrease in HHb as based on a mechanism known as neurovascular coupling.
Change in prefrontal cortex activation pattern through a fNIRS | during the intervention
  Analysis of Oxyhemoglobin (HbO2) and Deoxyhemoglobin (HHb) variation in four regions of interest (ROIs) in the PFC: left prefrontal dorsolateral cortex (LDLPFC); left medial prefrontal cortex (LMPFC); right medial prefrontal cortex (RMPFC); right dorsolateral prefrontal cortex (RDLPFC). An increase in brain activity is generally assumed to reflect an increase in HbO2 and decrease in HHb as based on a mechanism known as neurovascular coupling.

SECONDARY OUTCOMES:
Depressive symptomatology assessed through the Geriatric Depression Scale-15 (GDS-15) | baseline
  Participants' scores in the GDS-15. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 15 points. Higher scores indicate more severe depressive symptoms.
Change in depressive symptomatology assessed through the GDS-15 | 12 weeks after the beginning of the intervention
  Participants' scores in the GDS-15. This instrument evaluated depressive symptoms using yes/no answers. Scores range between 0 and 15 points. Higher scores indicate more severe depressive symptoms.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  Participants' answers in the sociodemographic questionnaire designed specifically for this study. It gathers information about gender, age, marital status, formal education, which social response the participant attends, medical comorbidities and cognitive symptoms and will be administered to all participants.
Adherence to the intervention and dropouts evaluated through a session form | during the intervention
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, regarding the attendance and mood/behavior of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; Rosa C Gomes Silva, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; Telmo A Santos Pereira, Ph.D., Principal Investigator — Polytechnic Institute of Coimbra, Coimbra Health School; João L Alves Apóstolo, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; Daniel F Borges Silva, M.Sc., Principal Investigator — Polytechnic Institute of Coimbra, Coimbra Health School
Locations (1):
- Cediara - Social Solidarity Association of Ribeira de Fráguas, Ribeira de Fráguas, Albergaria-a-Velha, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apóstolo JLA, Bobrowicz-Campos EM, dos Reis IAC, Henriques SJ, Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica. 2018; 23: 99-107. doi: 10.5944/rppc.vol.23.num.2.2018.21050
- [Background] Apóstolo J, Loureiro L, Reis I, Silva I, Cardoso D, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale -15 into Portuguese. Revista de Enfermagem Referência. 2014; IV(3): 65-73. doi: 10.12707/RIV14033
- [Background] Clare L, Woods RT. Cognitive training and cognitive rehabilitation for people with early-stage Alzheimer's disease: A review. Neuropsychological Rehabilitation. 2004; 14: 385-401. doi: 10.1080/09602010443000074
- [Background] Clare L, Wilson BA, Carter G, Breen K, Gosses A, Hodges JR. Intervening with everyday memory problems in dementia of Alzheimer type: an errorless learning approach. J Clin Exp Neuropsychol. 2000 Feb;22(1):132-46. doi: 10.1076/1380-3395(200002)22:1;1-8;FT132. PMID 10649552
- [Background] Davis RN, Massman PJ, Doody RS. Cognitive intervention in Alzheimer disease: a randomized placebo-controlled study. Alzheimer Dis Assoc Disord. 2001 Jan-Mar;15(1):1-9. doi: 10.1097/00002093-200101000-00001. PMID 11236819
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Filipin F, Feldman M, Taragano FE, Martelli M, Sánchez V, García V, et al. The efficacy of cognitive stimulation on depression and cognition in elderly patients with cognitive impairment: A retrospective cohort study. AIMS Medical Science. 2015; 3(1): 1-14. doi: 10.3934/medsci.2016.1.1
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia C. Adaptação à população portuguesa da tradução do Mini Mental State Examination. Revista Portuguesa de Neurologia. 1994; 1: 9-10.
- [Background] Justo-Henriques SI, Marques-Castro AE, Otero P, Vazquez FL, Torres AJ. [Long-term individual cognitive stimulation program in patients with mild neurocognitive disorder: a pilot study]. Rev Neurol. 2019 Apr 1;68(7):281-289. doi: 10.33588/rn.6807.2018321. Spanish. PMID 30906977
- [Background] Justo-Henriques SI, Otero P, Torres AJ, Vazquez FL. Effect of long-term individual cognitive stimulation intervention for people with mild neurocognitive disorder. Rev Neurol. 2021 Aug 15;73(4):121-129. doi: 10.33588/rn.7304.2021114. English, Spanish. PMID 34308545
- [Background] Lima CF, Meireles LP, Fonseca R, Castro SL, Garrett C. The Frontal Assessment Battery (FAB) in Parkinson's disease and correlations with formal measures of executive functioning. J Neurol. 2008 Nov;255(11):1756-61. doi: 10.1007/s00415-008-0024-6. Epub 2008 Sep 25. PMID 18821046
- [Background] Lobbia A, Carbone E, Faggian S, Gardini S, Piras F, Spector E, et al. The efficacy of cognitive stimulation therapy (CST) for people with mild-to-moderate dementia: A review. European Psychologist. 2018; 24(3): 257-277. doi: 10.1027/1016-9040/a000342
- [Background] Loewenstein DA, Acevedo A, Czaja SJ, Duara R. Cognitive rehabilitation of mildly impaired Alzheimer disease patients on cholinesterase inhibitors. Am J Geriatr Psychiatry. 2004 Jul-Aug;12(4):395-402. doi: 10.1176/appi.ajgp.12.4.395. PMID 15249277
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Novos valores normativos do Mini-Mental State Examination. Sinapse. 2009; 2: 10-16.
- [Background] Pereira T, Castro MA, Villafaina S, Carvalho Santos A, Fuentes-Garcia JP. Dynamics of the Prefrontal Cortex during Chess-Based Problem-Solving Tasks in Competition-Experienced Chess Players: An fNIR Study. Sensors (Basel). 2020 Jul 14;20(14):3917. doi: 10.3390/s20143917. PMID 32674476
- [Background] Verhulsdonk S, Hellen F, Hoft B, Supprian T, Lange-Asschenfeldt C. Attention and CERAD test performances in cognitively impaired elderly subjects. Acta Neurol Scand. 2015 Jun;131(6):364-71. doi: 10.1111/ane.12346. Epub 2014 Oct 28. PMID 25352352
- [Background] Wilson B. Towards a comprehensive model of cognitive rehabilitation. Neuropsychological Rehabilitation. 2002; 12(2): 97-110. doi: 10.1080/09602010244000020
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- See also: 2017 Demographic Statistics — https://www.ine.pt/xportal/xmain?xpid=INE&xpgid=ine_publicacoes&PUBLICACOESpub_boui=348174760&PUBLICACOESmodo=2
- See also: Dementia: assessment, management and support for people living with dementia and their carers — https://www.nice.org.uk/guidance/ng97/resources/dementia-assessment-management-and-support-for-people-living-with-dementia-and-their-carers-pdf-1837760199109
- See also: Mental health and older adults — http://www.who.int/mediacentre/factsheets/fs381/en/